CLINICAL TRIAL: NCT05579600
Title: Managed Care Updates of Subscriber Justice System Involvement for Suicide Prevention
Brief Title: Suicide Prevention for Justice Involved Managed Care Subscribers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1P50MH127512-01A1 8577; 1P50MH127512-01A1 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Suicide and Self-harm
Keywords: suicidal behavior; jail release; behavioral health providers; suicide training
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caring Contact letters (Experimental): Caring Contact letters will be mailed to a randomly selected group of managed care subscribers over a 6-month period following jail release.
  Interventions: Behavioral: Caring Contacts letters
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Caring Contacts letters — Caring Contacts involves sending individuals at risk for suicide brief, non- demanding messages of care.
  Arms: Caring Contact letters

SUMMARY:
The goal of this clinical trial is to test the effects of a suicide prevention intervention for individuals released from jail. The main question it aims to answer is: Does the use of Caring Contacts improve subscriber engagement with healthcare services while reducing suicide-related outcomes? Participants will include subscribers of a managed care organization (MCO). Intervention includes sending subscribers Caring Contacts letters for 6-months following jail release to target healthcare re-engagement and suicide prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Released from an Ohio jail
* enrolled in Medicaid through CareSource

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45155 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Arias, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arias SA, Sperber K, Jones R, Taxman FS, Miller TR, Zylberfuden S, Weinstock LM, Brown GK, Ahmedani B, Johnson JE. Managed care updates of subscriber jail release to prompt community suicide prevention: clinical trial protocol. BMC Health Serv Res. 2023 Nov 16;23(1):1265. doi: 10.1186/s12913-023-10249-5. PMID 37974126
- [Derived] Arias SA, Sperber K, Jones R, Taxman FS, Miller TR, Zylberfuden S, Weinstock LM, Brown GK, Ahmedani B, Johnson JE. Managed Care Updates of Subscriber Jail Release to Prompt Community Suicide Prevention: Clinical Trial Protocol. Res Sq [Preprint]. 2023 Sep 25:rs.3.rs-3350204. doi: 10.21203/rs.3.rs-3350204/v1. PMID 37841869

RESULTS

PARTICIPANT FLOW:
Groups:
- Caring Contact Letters: Caring Contacts involves sending individuals at risk for suicide brief, non-demanding messages of care.
- Caring Contact Control: No contact control condition for the Caring Contact letters
Period: Overall Study
Arm/Group | Caring Contact Letters | Caring Contact Control
Started | 22380 | 22775
Completed | 22380 | 22775
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caring Contact Letters | Caring Contact Control | Total
Number analyzed (Participants) | 22380 | 22775 | 45155
Age, Continuous [Mean (Standard Deviation); unit: Year] | 36.4 (10.9) | 36.4 (10.8) | 36.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8628 | 8702 | 17330
  Male | 13752 | 14073 | 27825
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Alaskan Native | 107 | 110 | 217
  Asian or Pacific Islander | 116 | 100 | 216
  Black (non-Hispanic) | 8528 | 8432 | 16960
  White (non-Hispanic) | 12746 | 13248 | 25994
  Hispanic | 25 | 28 | 53
  Native Hawaiian | 29 | 25 | 54
  Not Provided | 828 | 830 | 1658
  Other Race Ethnicity | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Suicide Attempt
Description: A suicide attempt is defined as "engaging in a potentially self-injurious behavior, associated with at least some intent to die as a result of the act." We will assess total number of subsequent attempts using the already-developed Mental Health Research Network (MHRN) algorithm for extracting suicide attempt information from claims data
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Number of suicide attempts
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of suicide attempts | .0202 (.3871) | .0229 (.5836)

2. Secondary Outcome: All-cause Injury and Poisoning
Description: All-cause injury and poisoning data will be extracted from ICD-10 data.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Number of all cause injury and poisoning
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of all cause injury and poisoning | 1.18 (3.74) | 1.17 (3.60)

3. Secondary Outcome: Outpatient Behavioral Health Service Linkage
Description: We will extract number of outpatient behavioral health (i.e., mental health or substance use) visits during the 12 months prior to and 6 months following jail release from claims data.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Number of behavioral health visits
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of behavioral health visits | 0.32 (4.96) | 0.34 (4.99)

4. Secondary Outcome: CareSource Member Services (CMS) Line Use
Description: Caring Contact messages will list the CMS phone number (which is answered by the Care Management Team, who are trained to assess and connect callers to the appropriate services) as a way to reach out. Care Source will track calls to this line by subscribers in all study conditions.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Number of calls
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of calls | 0.0088 (0.2284) | 0.0161 (1.3033)

5. Secondary Outcome: Inpatient and Emergency Department Mental Health Care Visits
Description: Data on inpatient and emergency department mental health visits will be extracted from claims data using MHRN algorithms.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of visits | 0.27 (1.55) | 0.28 (1.59)

6. Other Pre Specified Outcome: Number of Arrests
Description: We will also extract past year and next 6 month number of arrests from the Jail-Medicaid database.
Time Frame: 18 months
Measure: Number; unit: Number of arrests
Arm/Group | Caring Contact Letters | Caring Contact Control
Number analyzed (Participants) | 22380 | 22775
Number of arrests | 6355 | 6312

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 18 months
Arm/Group | Caring Contact Letters | Caring Contact Control
All-Cause Mortality (participants affected / at risk) | 0/22380 | 0/22775
Serious Adverse Events (participants affected / at risk) | 1177/22380 | 1071/22775
Other Adverse Events (participants affected / at risk) | 0/22380 | 0/22775
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caring Contact Letters (N=22380) | Caring Contact Control (N=22775)
Medically-treated Suicide Attempt (Psychiatric disorders) | 1177 | 1071
Inpatient hospitalization (potentially suicide-related) (Psychiatric disorders) | 1177 | 1071

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT05579600/Prot_SAP_000.pdf